CLINICAL TRIAL: NCT00404430
Title: Predictive Factors of Endothelial Function in Chronic Obstructive Disease Patients at the End of a Acute Exacerbation.
Brief Title: Protocol Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 0627
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Acute Respiratory Failure
Keywords: Endothelial function; Peripheral Arterial Tone; Systemic Inflammation; Oxidative Stress; Respiratory and peripheral muscular function; Cardiovascular risk; COPD severity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples for analysis of inflammatory and oxidative biological markers
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Exacerbated COPD patients: Patients with exacerbated COPD
- Stable COPD patients: Patients with stable COPD

SUMMARY:
The main objective of the study is to evaluate the predictive factors of the endothelial function to the waning of an acute exacerbation in COPD. It will act to do a multivariate analysis to determine the respective weight of the parameters of the systemic inflammation, of the oxidative stress of the functional respiratory parameters and then functional respiratory parameters.

In exacerbated Chronic Obstructive Pulmonary Disease (COPD) patients, there is augmentation of hypoxia and the obstructive ventilatory disorders is more important. This is correlated with an increase in C-reactive Protein (CRP) and of inflammatory cytokines and oxidative stress. It has been demonstrated that there is an endothelial dysfunction in answer to hypoxia. Since the exacerbated COPD patients are hypoxic in most cases , we suppose they have an endothelial dysfunction during exacerbation. So we think we will find an augmentation of vascular resistances ,shown by a peripheral arterial tone too high. And this, certainly, play a part in physiopathology of the COPD exacerbation.

DETAILED DESCRIPTION:
We want to judge the improvement of the endothelial function remotely to the acute exacerbation (6 weeks). And then we would like to correlate this improvement with the variations of oxidative stress, muscle strength, respiratory function and systemic inflammation.

We also would like to find a relation between the new hospitalizations for respiratory exacerbation and the initial value of endothelial function.

Then we would like to evaluate the relationship between the cardiovascular risk and the COPD severity.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with the waning of exacerbation:
* Male or Female more than 18 years old
* VEF1/FCV < 70% or COPD already knew
* At the moment of the respiratory failure, the day of the enter in hospital:
* Respiratory frequency >25
* PaCO2 > 45 mmHg
* pH < 7.35
* The day of the inclusion in our study:
* PH > 7.33 at the end of the respiratory failure, or 2 days of continuation, 3 to 7 days post acute exacerbation of continuation
* Fever < 38.5
* Patients who have signed the inform consent form
* Stable COPD patients:
* Men or women more than 18 years old
* VEF1/FCV < 70% or COPD already knew
* Patients who have signed the inform consent form

Exclusion Criteria:

* Evolutive obvious infection or CRP > 100 at inclusion Cardiac failure considered like the major cause of the exacerbation or cardiac insufficiency with FEVG < 45 %
* Smoker > 10 cigarettes a day Antioxidant catch: N-acetyl-cystein, selenium, ascorbic acid, alpha tocopherol acetate…
* Evolutive neoplasia
* Antioxidant catch: N-acetyl-cystein, selenium, ascorbic acid, alpha tocopherol acetate…
* pregnant women
* patient under supervision or trusteeship
* patient taking part in another clinical trial
* claustrophobia, patients allergic to contrast agents like Gadolinium, presence of material dissuading the realization of a MRI (pacemaker, implantable defibrillator, insulin pump, ferrometallic clips or foreign bodies in brain or eyes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with exacerbated (50) or stable (195) COPD
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2007-01-11 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
peripheral arterial tone | once a year

SECONDARY OUTCOMES:
Muscle strength measurements | once a year
biological markers of inflammation and oxidative stress | once a year
respiratory function measurements | once a year
Determine the relationship between the RMI measurements and the cardiovascular risk | once during the study
Determine the relationship between the hospitalizations for decompensation and the initial value of endothelial function | study time frame
Determine the relationship between the RMI measurements and the COPD severity | once during the study
Determine the prevalence of nocturnal non-dipping blood pressure in COPD patients | once a year

OTHER OUTCOMES:
pulse wave velocity measurement | once a year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis JP Pépin, ProfessorPhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- France : Laboratoire EFCR - Functional Cardio-Respiratory Exploration Laboratory, Grenoble, Isere, France

REFERENCES:
- [Background] Malo O, Sauleda J, Busquets X, Miralles C, Agusti AG, Noguera A. [Systemic inflammation during exacerbations of chronic obstructive pulmonary disease]. Arch Bronconeumol. 2002 Apr;38(4):172-6. Spanish. PMID 11953269
- [Background] Vassilakopoulos T, Katsaounou P, Karatza MH, Kollintza A, Zakynthinos S, Roussos C. Strenuous resistive breathing induces plasma cytokines: role of antioxidants and monocytes. Am J Respir Crit Care Med. 2002 Dec 15;166(12 Pt 1):1572-8. doi: 10.1164/rccm.200203-177OC. Epub 2002 Oct 3. PMID 12406849
- [Background] Yende S, Waterer GW, Tolley EA, Newman AB, Bauer DC, Taaffe DR, Jensen R, Crapo R, Rubin S, Nevitt M, Simonsick EM, Satterfield S, Harris T, Kritchevsky SB. Inflammatory markers are associated with ventilatory limitation and muscle dysfunction in obstructive lung disease in well functioning elderly subjects. Thorax. 2006 Jan;61(1):10-6. doi: 10.1136/thx.2004.034181. Epub 2005 Nov 11. PMID 16284220
- [Background] Barreiro E, de la Puente B, Minguella J, Corominas JM, Serrano S, Hussain SN, Gea J. Oxidative stress and respiratory muscle dysfunction in severe chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 May 15;171(10):1116-24. doi: 10.1164/rccm.200407-887OC. Epub 2005 Feb 25. PMID 15735057
- [Background] Lerman A, Zeiher AM. Endothelial function: cardiac events. Circulation. 2005 Jan 25;111(3):363-8. doi: 10.1161/01.CIR.0000153339.27064.14. No abstract available. PMID 15668353
- [Result] Mallia P, Johnston SL. Mechanisms and experimental models of chronic obstructive pulmonary disease exacerbations. Proc Am Thorac Soc. 2005;2(4):361-6; discussion 371-2. doi: 10.1513/pats.200504-025SR. PMID 16267363
- [Derived] Minet C, Vivodtzev I, Tamisier R, Arbib F, Wuyam B, Timsit JF, Monneret D, Borel JC, Baguet JP, Levy P, Pepin JL. Reduced six-minute walking distance, high fat-free-mass index and hypercapnia are associated with endothelial dysfunction in COPD. Respir Physiol Neurobiol. 2012 Aug 15;183(2):128-34. doi: 10.1016/j.resp.2012.06.017. Epub 2012 Jun 18. PMID 22721944
- [Derived] Vivodtzev I, Minet C, Wuyam B, Borel JC, Vottero G, Monneret D, Baguet JP, Levy P, Pepin JL. Significant improvement in arterial stiffness after endurance training in patients with COPD. Chest. 2010 Mar;137(3):585-92. doi: 10.1378/chest.09-1437. Epub 2009 Oct 31. PMID 19880908